CLINICAL TRIAL: NCT00817947
Title: An Assessment of the Short-Term Effects of the Airway Clearance Technique of High Frequency Chest Wall Oscillation in People With Cystic Fibrosis
Brief Title: Airway Clearance Using High Frequency Chest Wall Oscillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Dr Jennifer A Pryor, Royal Brompton & Harefield NHS Trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q0404/54
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Cystic Fibrosis
Keywords: Airway clearance; Cystic fibrosis; High frequency chest wall oscillation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual airway clearance technique (Active Comparator): Airway clearance using the active cycle of breathing techniques, autogenic drainage, positive expiratory pressure or oscillating positive expiratory pressure
  Interventions: Device: High frequency chest wall oscillation
- HFCWO (Other): High frequency chest wall oscillation
  Interventions: Device: High frequency chest wall oscillation

INTERVENTIONS:
Device: High frequency chest wall oscillation — Airway clearance using high frequency chest wall oscillation ('The Vest')

SUMMARY:
High frequency chest wall oscillation (HFCWO) has been shown to increase tracheal mucous clearance compared with control. These observations led to the development of 'The Vest' which is a non-stretchable jacket connected to an air-pulse generator and worn by the patient over the chest wall. The generator rapidly inflates and deflates 'The Vest' which gently compresses and releases the chest wall between 5 and 20 times per second. This generates mini-coughs which are said to dislodge mucus from the bronchial walls and to facilitate its movement up the airways. In addition 'The Vest' has been shown to reduce the viscosity of mucus and this should further enhance mucous clearance. The technique has, for many years, been widely used in the United States of America as an alternative to the European airway clearance regimens of the active cycle of breathing techniques, autogenic drainage, positive expiratory pressure and oscillating positive expiratory pressure, but 'The Vest' has only recently been registered for use in Europe. It is important that the airway clearance regimen of 'The Vest' be compared with the alternative airway clearance regimens widely used in Europe.

Hypothesis: In people with cystic fibrosis 'The Vest' will lead to the expectoration of an increased weight of sputum during treatment sessions compared with alternative airway clearance regimens.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cystic fibrosis
* 16 years of age or over
* forced expiratory volume in one second greater than or equal to 25 percent of predicted
* hospitalised patients in a stable clinical state

Exclusion Criteria:

* current severe haemoptysis
* rib fractures
* pregnancy
* inability to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Weight of sputum expectorated | Twenty-four hours

SECONDARY OUTCOMES:
Forced expiratory volume in one second | One hour (before and 30 minutes after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Pryor, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom